CLINICAL TRIAL: NCT01160627
Title: Prevention of Contrast-induced Nephropathy in Patients With Acute Myocardial Infarction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Lisette Okkels Jensen, MD DMSci PhD, Odense University Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CIN in STEMI
Record Dates: First submitted 2010-07-09; First posted 2010-07-12 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Contrast Induced Nephropathy
Keywords: CIN STEMI
MeSH Terms: interventions — Acetylcysteine; Sodium Bicarbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Standard treatment (Active Comparator): Hydration
  Interventions: Other: Hydration
- Combined Acetylcystein and Sodium Bicarbonat (Active Comparator)
  Interventions: Drug: Combined Acetylcystein and Sodium Bicarbonate
- Sodium Bicarbonate (Active Comparator)
  Interventions: Drug: Sodium bicarbonate
- Acetylcystein for 2 days (Active Comparator): Standard treatment + acetylcystein for 2 days
  Interventions: Drug: Acetylcysteine

INTERVENTIONS:
Other: Hydration — Saline hydration
  Arms: Standard treatment
Drug: Acetylcysteine — Acetylcystein tablets for 2 days
  Arms: Acetylcystein for 2 days
Drug: Sodium bicarbonate — Sodium bicarbonate 500 ml followed by 100 ml/hour for 5 hours
  Arms: Sodium Bicarbonate
Drug: Combined Acetylcystein and Sodium Bicarbonate — Sodium bicarbonate 500 ml followed by 100 ml/hour for 5 hours combined with acetylcystein tablets for 2 days
  Arms: Combined Acetylcystein and Sodium Bicarbonat

SUMMARY:
OBJECTIVE: To evaluate the efficacy of prevention of contrast induced nephropathy in patients with ST segment elevation myocardial infarction treated with primary percutaneous coronary intervention.

DESIGN: Prospective study. SETTING: Three-center study Acute kidney injury was defined as a rise in creatinine >25% from baseline Serum creatinine will be measured at baseline and each day for the following 3 days and at 30 days.

Patients will be randomised to:

1. Standard treatment
2. Standard treatment + acetylcystein for 2 days
3. Standard treatment + Sodium bicarbonate 500 ml / followed by 100 ml/h for 5 hours
4. Standard treatment + acetylcystein for 2 days + Sodium bicarbonate 500 ml / followed by 100 ml/h for 5 hours

ELIGIBILITY:
Inclusion Criteria:

* STEMI patients treated with primary PCI

Exclusion Criteria:

* Cardiogenic shock

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Actual)
Dates: Start 2010-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Prevention of contrast induced nephropathy in STEMI patients treated with primary PCI | from baseline to day 3
  Rise in creatinine >25% from baseline to day 3

SECONDARY OUTCOMES:
Prevention of contrast induced nephropathy in STEMI patients treated with primary PCI | from baseline to day 30
  Rise in creatinine >25% from baseline to day 30

CONTACTS AND LOCATIONS:
Overall Officials: Per Thayssen, MD DMSci, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

REFERENCES:
- [Derived] Thayssen P, Lassen JF, Jensen SE, Hansen KN, Hansen HS, Christiansen EH, Junker A, Ravkilde J, Thuesen L, Veien KT, Jensen LO. Prevention of contrast-induced nephropathy with N-acetylcysteine or sodium bicarbonate in patients with ST-segment-myocardial infarction: a prospective, randomized, open-labeled trial. Circ Cardiovasc Interv. 2014 Apr;7(2):216-24. doi: 10.1161/CIRCINTERVENTIONS.113.000653. Epub 2014 Apr 8. PMID 24714489